CLINICAL TRIAL: NCT07129876
Title: Effects of Simulator Motion Fidelity on Pilot Performance While Using a Mixed-Reality Headset
Brief Title: Motion Fidelity Effects With Mixed-Reality
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Aeronautics and Space Administration (NASA) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: STUDY00000883
Record Dates: First submitted 2025-06-05; First posted 2025-08-19 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Simulator Motion Variations (Experimental): 2 flight tasks; 4 motion conditions; 3 repetitions per condition (n = 12 per task)
  Interventions: Other: Simulator Motion

INTERVENTIONS:
Other: Simulator Motion — Motion fidelity of the simulator.

SUMMARY:
The purpose of this research is to investigate how different levels of simulator motion fidelity affect pilot performance in two different flight tasks while using a head mounted display (or mixed-reality headset) for out-the-window (OTW) visuals. Three levels of motion fidelity will be studied: 1) no motion, 2) small hexapod motion, and 3) one-to-one vehicle motion.

DETAILED DESCRIPTION:
The aim of this study is to determine the effects of simulator motion fidelity on pilot performance in two demanding piloting tasks while wearing a mixed-reality headset for OTW visuals. Pilots will be exposed to mixed-reality visuals meaning that the virtual OTW visual scene will be overlayed on an image of the real simulator cockpit and head down displays (HDD). Pilots will fly two tasks in this experiment: 1) a roll-lateral sidestep maneuver, and 2) a precision landing.

In task 1, the roll-lateral sidestep maneuver will be from one landing pad to a second landing pad of a vertiport on the Fifth & Mission Parking Garage in San Francisco. The vertiport is in a San Francisco visual database surrounded by buildings with high-resolution textures. Pilots are instructed to stay at a constant altitude. A positioning sight will be placed in the visual scene at each landing pad to allow pilots to determine their positioning error precisely. Pilots will be provided with lateral position and time criteria for desired and adequate performance. Pilots will be instructed to press an event marker on their control inceptor when they acquire the station-keeping point at the landing pad. Turbulence will be used to make the task more difficult. This task will be similar to the roll-lateral experiment described by Schroeder that was also performed in the VMS.

In task 2, pilots will perform a landing at the same vertiport in San Francisco that is used in task 1. The task will start from level flight from a position that allows for a standard approach and landing. Landing position and time criteria for desired and adequate performance will be communicated to the pilots. Pilots will press an event marker on the control inceptor when they acquire the desired reference point on the landing pad. Turbulence will be introduced to make the task more difficult.

Pilots will receive the informed consent form and a Motion Sickness Susceptibility Questionnaire (MSSQ via email first. They will be asked to fill out the MSSQ at home and return it to the PI before being scheduled and coming to the VMS. On the day of the experiment, participants will first receive a briefing and walkaround of the facility before providing their informed consent (60 minutes). Next, they will take a seat in the simulator cab where seat and headset adjustments will be made first to make sure the experiment can be performed comfortably. This is followed by the first data-collection session in which one of the tasks is flown (45 minutes). Both tasks will be flown under three motion fidelity conditions described in Section 8.3 below. Three repetitions of each motion condition will be flown for both tasks, after completing three training runs, for a total of 12 runs per task. A 30-minute break is scheduled after the first data-collection session. The second session in which the other tasks is flown will commence after the break (45 minutes). Finally, pilots will be debriefed and can ask any remaining questions (30 minutes).

Pilot performance in each task will be determined by several outcome-based variables, including the error between desired and actual aircraft position and attitude at specified locations, the intensity of control inputs, and task completion time. Pilots will also complete a motion fidelity rating and a Simulator Sickness Questionnaire (SSQ) at the end of each run.

Hypothesis: Pilot performance and subjective motion ratings will be significantly different between the different simulator motion fidelity conditions.

Before data analysis, all data will be averaged over the three repetitions of each condition. A one-way repeated-measures Multivariate Analysis of Variance (MANOVA) will be used on the data from each task to determine statistically significant effects. If test assumptions are not met (e.g., homogeneity of covariance matrices), corrections or appropriate alternate tests will be used. Any reporting of the statistical results will include the F statistic (or equivalent for alternate tests), degrees of freedom, probability values, and effect sizes.

Based on previous studies investigating the effects of motion fidelity on pilot performance, it is expected that pilot performance will be lower without simulator motion or with small-hexapod motion compared to one-to-one vehicle motion. Control intensity will show the opposite trend; that is, will be higher without simulator motion and will decrease with higher motion fidelity.

ELIGIBILITY:
Inclusion Criteria:

* Normal or corrected to normal vision.

Exclusion Criteria:

* Claustrophobia.
* Susceptible to motion sickness.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2025-05-19 (Actual); Primary Completion 2025-05-30 (Actual); Study Completion 2025-05-30 (Actual)

PRIMARY OUTCOMES:
Time to Complete Flight Task Maneuver (Averaged over Repetitions) | Day 1
  Time needed to complete (a portion of) the flight task measured against desired and adequate performance criteria:
  Heliport Approach Task - Battery time remaining (desired >=20:00 min, adequate >=19:40 min)
  Lateral Reposition and Hold Task
  - Reposition completion time (desired <=25 s, adequate <=35 s)
Accuracy of the Flight Task Maneuver (Averaged over Repetitions) | Day 1
  Accuracy of the maneuver during (a portion of) the flight task measured against desired and adequate performance criteria:
  Heliport Approach Task
  * Glideslope deviation (desired +-0.7 deg, adequate +-2.1 deg)
  * Localizer deviation (desired +-0.7 deg, adequate +-2.1 deg)
  * Helipad boundary crossing height (desired +-10 ft, adequate +-20 ft)
  * Helipad boundary crossing speed (desired +-5 kts, adequate +-10 kts)
  * Helipad center deviation (desired +-20 ft, adequate +-60 ft)
  Lateral Reposition and Hold Task
  * Ground track deviation (desired +-5 ft, adequate +-10 ft)
  * Target ground speed deviation (desired +-5 kts, adequate +-8 kts)
  * Altitude deviation (desired +-5 ft, adequate +-10 ft)
  * Heading deviation (desired +-10 deg, adequate +-15 deg)
  * Hover point lateral and longitudinal deviation (desired +-5 ft, adequate +-10 ft)
Motion Fidelity Rating | Day 1
  Possible answers are: Low Fidelity, Medium Fidelity, High Fidelity

SECONDARY OUTCOMES:
Simulator Sickness Questionnaire (SSQ) | Day 1
  This questionnaire requires rating 16 symptoms with a scale from none, slight, moderate, to severe. The symptoms are: general discomfort, fatigue, headache, eye strain, difficulty focusing, increased salivation, sweating, nausea, difficulty concentrating, fullness of head, blurred vision, dizzy (eyes open), dizzy (eyes closed), vertigo, stomach awareness, burping.

CONTACTS AND LOCATIONS:
Locations (1):
- NASA Ames Research Center, Vertical Motion Simulator, Mountain View, California, United States

IPD SHARING:
Plan to Share IPD: No